CLINICAL TRIAL: NCT03271749
Title: Protocol for Accelerated Recovery in Patients Undergoing Thoracic Surgical Procedures Adapted to the Conditions of Santa Marcelina - Itaquera Hospital - São Paulo - Brazil (PROSM). Study Randomized Comparative Between the Adoption of the Proposed Guidelines and the Traditional Method Currently Used in the Institution
Brief Title: Protocol for Accelerated Recovery in Patients Undergoing Thoracic Surgical Procedures (PROSM). Study Randomized Comparative Between the Adoption of the Proposed Guidelines and the Traditional Method Currently Used in the Institution
Acronym: PROSM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Igor Renato Louro Bruno de Abreu (Other)
Responsible Party: Sponsor-Investigator, Igor Renato Louro Bruno de Abreu, Assistant physician of the thoracic surgery team of the Hospital Santa Marcelina de Itaquera, Hospital Santa Marcelina
Organization: Hospital Santa Marcelina (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 70142917.0.0000.0066
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Pain; Postoperative Complications; Postoperative Nausea; Lung Cancer
Keywords: Fast Track surgical recovery; Surgical recovery; Thoracic surgery
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications; Postoperative Nausea and Vomiting; Lung Neoplasms | interventions — Anesthesia; Postoperative Care

STUDY DESIGN:
Intervention Model Description: Randomized controlled Trial
Who Masked: Outcomes Assessor
Masking Description: It's impossible to mask the participants, care providers and investigators, because of the apparent differences in both techniques. For this reason the data analysis will be masked to avoid influences by the other participants during the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (No Intervention): The participants of this arm will receive the convencional pre operative, anesthesia and postoperative care for lung resections for treatment of lung neoplasms
- PROSM interventional (Experimental): The participants of this arm will receive the PROSM protocol pre operative, anesthesia and postoperative care for lung resections for treatment of lung neoplasms
  Interventions: Other: PROSM guidelines for preoperative, anesthesia and postoperative care for lung resections

INTERVENTIONS:
Other: PROSM guidelines for preoperative, anesthesia and postoperative care for lung resections — The PROSM guidelines is described previously in study description
  Arms: PROSM interventional

SUMMARY:
Introduction:

Aiming at reducing costs and optimizing the use of these financial resources, several postoperative recovery protocols have emerged that aim to reduce the length of hospital stay by accelerating surgical recovery.1,2 In view of the current Brazilian political and economic scenario allied to the existing scientific knowledge on the subject , the investigators developed a protocol that aims to meet this need using resources already available and offered in brazilian public health system. The investigators called this protocol as Protocol of Operative Recovery Santa Marcelina (PROSM) that had as inspiration the protocols of accelerated postoperative recovery already used in several European health services.

Goals:

1. To evaluate the impact of PROSM on the length of hospitalization in days and postoperative pain (visual analog pain scale - VAS) in patients submitted to surgical procedures performed by the thoracic surgery team of the Hospital Santa Marcelina de Itaquera.
2. Evaluate the impacts of PROSM in reducing the costs (US dollars) of surgical treatment and hospitalization of these patients.

Materials and methods:

A group of 200 patients with elective pulmonary resections (segmentectomies, lobectomies or pneumonectomies) to treat neoplastic lung diseases will be selected by the investigators.

The participants will be randomized into two groups (rate of randomization 1/1).

The first group will be submitted to the standard surgical treatment that is currently used in Santa Marcelina - Itaquera hospital. The second group will be submitted to treatment with the adoption of the PROSM guidelines, which will be detailed later.

Investigators will evaluate in the two groups: surgical time in minutes, intraoperative complications: intraoperative bleeding in mililiters, need for transfusion of blood products, intraoperative clinical complications. Investigators will also evaluate the need for postoperative recovery in Intensive Care Unit (ICU), medications used to maintain the anesthetic plane during the procedure (amount of drugs in milligrams), medications used for postoperative analgesia, length of hospital stay in days, postoperative clinical complications, need for surgical re-boarding, immediate postoperative pain (VAS), postoperative pain at the time of discharge and the first outpatient return (VAS), the need for opioid analgesics at home after discharge.

After the data collection, the investigators will analyze them and make a comparative study of the costs of surgical treatment and hospitalization between the two groups. This data will be obtained from the billing department of the Hospital Santa Marcelina de Itaquera.

DETAILED DESCRIPTION:
Introduction:

Patients submitted to surgical procedures for the treatment of thoracic diseases, whether benign or neoplastic, are exposed to potential complications.

The main complications related to these procedures are primarily lung infections, followed by thrombotic events, cardiovascular events, and complications due to previous chronic diseases.

Faced with the occurrence of complications, these patients require a longer hospitalization period, using high cost medications, generating additional unexpected costs.

Aiming at reducing costs and optimizing the use of these financial resources, several postoperative recovery protocols have emerged that aim to reduce the length of hospital stay by accelerating surgical recovery.1,2 In view of the current Brazilian political and economic scenario allied to the existing scientific knowledge on the subject , the investigators developed a protocol that aims to meet this need using resources already available and offered in brazilian public health system. The investigators called this protocol as Protocol of Operative Recovery Santa Marcelina (PROSM) that had as inspiration the protocols of accelerated postoperative recovery already used in several European health services.

Goals:

1. To evaluate the impact of PROSM on the length of hospitalization in days and postoperative pain (visual analog pain scale - VAS) in patients submitted to surgical procedures performed by the thoracic surgery team of the Hospital Santa Marcelina de Itaquera.
2. Evaluate the impacts of PROSM in reducing the costs (US dollars) of surgical treatment and hospitalization of these patients.

Materials and methods:

A group of 200 patients with elective pulmonary resections (segmentectomies, lobectomies or pneumonectomies) to treat neoplastic lung diseases will be selected by the investigators.

Patients under the age of eighteen years old, unable to read, understand and sign informed consent, patients with compromised performance status (ECOG greater than 2), patients with a body mass below 60 kilograms or greater than 120 kilograms , patients with allergy to latex, patients with a history of allergy to any of the drugs used in anesthesia for PROSM, patients with renal dysfunction, liver dysfunction and severe cardiac dysfunction (cardiac failure), will be excluded from this study.

The participants will be randomized into two groups (rate of randomization 1/1). The first group will be submitted to the standard surgical treatment that is currently used in Santa Marcelina - Itaquera hospital. The second group will be submitted to treatment with the adoption of the PROSM guidelines, which will be detailed later.

Investigators will evaluate in the two groups: surgical time in minutes, intraoperative complications: intraoperative bleeding in mililiters, need for transfusion of blood products, intraoperative clinical complications. Investigators will also evaluate the need for postoperative recovery in Intensive Care Unit (ICU), medications used to maintain the anesthetic plane during the procedure (amount of drugs in milligrams), medications used for postoperative analgesia, length of hospital stay in days, postoperative clinical complications, need for surgical re-boarding, immediate postoperative pain (VAS), postoperative pain at the time of discharge and the first outpatient return (VAS), the need for opioid analgesics at home after discharge. The follow-up time of these patients for the purpose of collecting data for this study will be started with their agreement to participate in the project and with the signing of the free and informed consent term and will extend until the third postoperative return. After this period, the participants will be followed for assistance purposes only.

After the data collection, this will be analyzed and a comparative study of the costs of surgical treatment and hospitalization between the two groups will be made. This data will be obtained from the billing department of the Santa Marcelina - Itaquera hospital.

Continuous variables will be expressed as medians with deviations. Categorical variables will be represented by absolute numbers and percentages. The Gaussian distribution of the variables will be tested using Kolmogorov - Smirnov test. The comparison between medians will be evaluated through the use of Student's T test. The comparison between categorical variables will be carried out using Chi-square test. Possible risk factors that contribute to an increase in the length of hospital stay and an increase in postoperative pain will be traced through the use of logistic regressions.

The analysis of the data will be carried out using the software Statistical Package for the Social Sciences (SPSS) 17.0 software (SPSS, Chicago, IL, USA)

PROSM Guidelines Description:

Selected patients who agree to participate in the present project and whose randomization assign them to the intervention PROSM group will be submitted to the following guidelines.

Preoperative care: In addition to conventional preoperative care including cessation of smoking and use of medications for comorbidities treatment, guidelines for preoperative fasting, verification of preoperative exams and cardiovascular and pre-anesthetic evaluations, the patient will receive guidelines for home exercises to perform daily walks with thirty minutes duration until the day of surgery. This measure aims to create in the patient the habit of moving daily. This will facilitate adherence to the proposed exercises for postoperative recovery.

On the day of surgery, immediately before the patient is taken to the operating room, we will administer 8 drops of chlorpromazine solution and 750 milligrams of paracetamol or 500 milligrams of dipyrone. The goal is to generate preemptive analgesia. Patients who admitted to the surgical procedure exhibit evidence of abandonment of the preoperative guidelines will be excluded from the study.

Anesthesia: The participant will be adequately monitored with pulse oximetry, cardioscopy, capnography, noninvasive blood pressure, temperature monitoring, anesthetic depth monitoring through the BIS method (bispectral index), delayed bladder catheter. The necessity or not of central venous access and invasive blood pressure will be evaluated according to the cardiovascular risks and the size of the surgery. For pulmonary resection operations we will use selective orotracheal intubation as already agreed in the institution.

Anesthetic induction will be performed using short duration opioid (remifentanil), hypnotic (propofol) and neuromuscular blocker with dose adjusted according to the patient's body mass.3 Intraoperative analgesia will be obtained through paravertebral and incisional intercostal block through the infiltration of a drug solution containing 500mililiters of saline, 1 vial of 5milligrams / 20milliliters bupivacaine, 20milliliters of lidocaine 2% without vasoconstrictor, 10milligrams of dexamethasone , 500milligrams of hydrocortisone, 75milligrams of clonidine, 5milligrams of ketamine and 40milliliters of sodium bicarbonate 8.4% solution). Investigators will use only the volume of solution sufficient to generate the intercostal blocks of the spaces pertaining to the incision and the orifice of the pleural drain and completely infiltrate the surgical wound. The surplus drug solution will be discarded.4 The participants will not be submitted to epidural anesthesia, only to the block.

Intercostal block and infiltration of the surgical wound will be performed by the surgical team while the other anesthetic procedures will be performed and accompanied by the anesthesiologist. At any time during the procedure, the anesthesiologist may administer additional anesthetic drugs or any other type of drug deemed necessary to ensure adequate pain control and hemodynamic stability of the patient. Throughout the procedure there should be dialogue and exchange of information between the surgical and anesthetic teams.

Anesthetic recovery: Post anesthetic recovery will commence immediately after the surgical dressing. The participants will be placed in horizontal dorsal decubitus, the anesthetic drugs will be switched off, the patient will receive intravenous antiemetic (ondansetron) and intravenous non-steroidal anti-inflammatory drug (ketoprofen) before extubation to avoid nausea and decrease postoperative pain. The patient will be extubated as soon as he is recovering his consciousness and is able to maintain an effective spontaneous breath.

Immediately after the extubation, the surgeon will elevate the decubitus of the surgical table to 45 degrees maintaining the constant observation of the blood pressure, heart rate and pulse oximetry. It will remain elevated until the patient is well awake. If the patient is unable to maintain a sufficient level of consciousness to understand and respond to verbal commands within 50 minutes of extubation or if during awakening the patient develops postural hypotension surgical team will abort the protocol and resume recovery by conventional measures.5 These cases will be counted as failure to execute the method.

When the patient is conscious and able to understand sentences and respond to verbal commands, investigators will begin the postoperative exercise program. Initially participant will do breathing exercises with inspirations and forced exhalations followed by elevation and lowering of the upper limbs.

While the participant is in the operating room, sequences of 10 exercises with a 1-minute interval between sequences will be performed.5 From the moment the anesthesiologist authorizes, the patient will be referred for anesthetic recovery room Upon reaching anesthetic recovery room, the patient will receive water and diet. After feeding, will be placed in an armchair, maintaining monitoring where will continue to do breathing exercises, lifting and lowering exercises of the upper limbs and extension and flexion of lower limbs. At this moment the participant will be accompanied by a doctor of the surgical team and a physiotherapist who will guide him in relation to the movements. A family escort will be allowed to remain with the patient helping to do the exercises. This phase of recovery will last 2 hours.5, 6 After this period of time, the physician representing the surgical team will put the patient on stand and watch the patient for 4 minutes in order to evaluate possible postural hypotension and assess the patient's ability to support his or her own weight. If the patient does not tolerate standing, participant will be placed back in the armchair and will continue with the exercises. Otherwise, the physician and physiotherapist will walk with the patient into the anesthetic recovery room for a period of 30 minutes with rest breaks as needed.

Referral to the hospitalization unit: After anesthesia recovery, the participants will be referred to the hospitalization units. In the hospitalization units the patient will do a 15 minute walk in the hallway every 60 minutes interval. During the intervals the patient will be resting in an armchair doing the movements previously described.

Those patients at risk of postoperative cardiac arrhythmias who received intraoperative blood products with a risk for hemorrhagic events using some type of vasoactive drug requiring ventilatory support will be referred to the ICU where they will remain for at least 24 hours , maintaining the same lines of proposed postoperative exercises. Indication or not of ICU postoperatively should be a consensus between surgical team and anesthetic team.7

Postoperative Prescription: The postoperative prescription should contain a general voluntary diet, medications that the patient already use, prophylactic antibiotics in the first 24 hours of the postoperative period, dipyrone or paracetamol of schedule, ketoprofen of schedule or toragesic, methadon 5milligrams per mouth if pain, antiemetics (ondansetron) schedule, laxative once a day, chlorpromazine solution drops (from 8 to 10 drops) at nigth. Investigators should not prescribe anticoagulants or antiplatelet agents until the patient has 7 days postoperative. There is no need for prophylactic enoxaheparin because the patient will be in continuous movement. Daily radiographs will be performed while the patient has a thoracic drainage. Laboratory tests will be requested only if the patient shows some type of abnormality on the physical examination that raises some suspicion of organic dysfunction or if there is any indication for it based on the preoperative cardiovascular and anesthetic evaluations.

Discharge: When the patient is in conditions for hospital discharge, this will be done through some guidelines:

1. Return to the outpatient thoracic surgery in 7 days to continue postoperative follow-up.
2. Prescription of analgesics for home use.
3. Guidance on possible postoperative complications, making it very clear in which circumstances the patient should return to the emergency room (fever, dyspnea, bleeding or chest pain refractory to the use of medication).

ELIGIBILITY:
Inclusion Criteria:

* patients with elective pulmonary resections (segmentectomies, lobectomies or pneumonectomies) to treat neoplastic lung diseases.

Exclusion Criteria:

* unable to read, understand and sign informed consent
* patients with compromised performance status (ECOG greater than 2)
* body mass below 60 kg or greater than 120 kg
* allergy to latex
* patients with a history of allergy to any of the drugs used in anesthesia for PROSM
* patients with renal dysfunction
* liver dysfunction
* severe cardiac dysfunction (cardiac failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
length of hospitalization in days | 1825 days
  To evaluate the impact of PROSM on the length of hospitalization in patients submitted to surgical procedures by thoracic surgery team of the Santa Marcelina - Itaquera hospital
postoperative pain using visual analog pain scale (VAS) | 1825 days
  To evaluate the impact of PROSM on postoperative pain in patients submitted to surgical procedures by thoracic surgery team of the Santa Marcelina - Itaquera hospital

SECONDARY OUTCOMES:
costs of surgical treatment in US dollars | 1825 days
  Evaluate the impacts of PROSM in reducing the costs of surgical treatment and hospitalization of these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando C Abrão, M.D., Study Chair — Coordinating physician of the thoracic surgery team of Santa Marcelina de Itaquera Hospital
Locations (1):
- Ambulatório de Nódulos e Massas Pulmonares H Santa Marcelina, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
We are planning to publish partial data analysis during the study period

REFERENCES:
- [Background] Dong Q, Zhang K, Cao S, Cui J. Fast-track surgery versus conventional perioperative management of lung cancer-associated pneumonectomy: a randomized controlled clinical trial. World J Surg Oncol. 2017 Jan 13;15(1):20. doi: 10.1186/s12957-016-1072-5. PMID 28086896
- [Background] Wolk S, Meissner T, Linke S, Mussle B, Wierick A, Bogner A, Sturm D, Rahbari NN, Distler M, Weitz J, Welsch T. Use of activity tracking in major visceral surgery-the Enhanced Perioperative Mobilization (EPM) trial: study protocol for a randomized controlled trial. Trials. 2017 Feb 21;18(1):77. doi: 10.1186/s13063-017-1782-1. PMID 28222805
- [Background] Jones NL, Edmonds L, Ghosh S, Klein AA. A review of enhanced recovery for thoracic anaesthesia and surgery. Anaesthesia. 2013 Feb;68(2):179-89. doi: 10.1111/anae.12067. Epub 2012 Nov 5. PMID 23121400
- [Background] Komatsu T, Kino A, Inoue M, Sowa T, Takahashi K, Fujinaga T. Paravertebral block for video-assisted thoracoscopic surgery: analgesic effectiveness and role in fast-track surgery. Int J Surg. 2014;12(9):936-9. doi: 10.1016/j.ijsu.2014.07.272. Epub 2014 Aug 1. PMID 25091399
- [Background] Das-Neves-Pereira JC, Bagan P, Coimbra-Israel AP, Grimaillof-Junior A, Cesar-Lopez G, Milanez-de-Campos JR, Riquet M, Biscegli-Jatene F. Fast-track rehabilitation for lung cancer lobectomy: a five-year experience. Eur J Cardiothorac Surg. 2009 Aug;36(2):383-91; discussion 391-2. doi: 10.1016/j.ejcts.2009.02.020. Epub 2009 Mar 26. PMID 19324571
- [Background] Chen L, Sun L, Lang Y, Wu J, Yao L, Ning J, Zhang J, Xu S. Fast-track surgery improves postoperative clinical recovery and cellular and humoral immunity after esophagectomy for esophageal cancer. BMC Cancer. 2016 Jul 11;16:449. doi: 10.1186/s12885-016-2506-8. PMID 27401305
- [Background] Asteriou C, Lazopoulos A, Rallis T, Gogakos AS, Paliouras D, Barbetakis N. Fast-track rehabilitation following video-assisted pulmonary sublobar wedge resection: A prospective randomized study. J Minim Access Surg. 2016 Jul-Sep;12(3):209-13. doi: 10.4103/0972-9941.183483. PMID 27279390